CLINICAL TRIAL: NCT06887712
Title: Efficacy of Oral Midazolam for Sedation and Amnesia in Preschool Children Undergoing Dental Procedures: a Randomized Controlled Trial
Brief Title: Efficacy of Oral Midazolam for Sedation and Amnesia in Preschool Children Undergoing Dental Procedures
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: Hanoi national hospital of odonto stomatology (Unknown)
Responsible Party: Principal Investigator, DUC NGUYEN MINH, Lecturer, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCSPQKRHM
Record Dates: First submitted 2025-03-16; First posted 2025-03-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2023-06

CONDITIONS: Dental Anxiety
Keywords: Oral Midazolam; Sedation; Amnesia; Pediatric Dentistry,
MeSH Terms: conditions — Amnesia | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Oral Midazolam 0.3 mg/kg (Experimental): Arm 1: Oral Midazolam 0.3 mg/kg Children aged 3-6 years with dental anxiety receive oral midazolam at a dose of 0.3 mg/kg prior to dental procedures. Sedative and amnesic effects, patient cooperation, and safety outcomes are evaluated.
  Interventions: Drug: Oral midazolam
- Arm 2: Oral Midazolam 0.6 mg/kg (Experimental): Arm 2: Oral Midazolam 0.6 mg/kg Children aged 3-6 years with dental anxiety receive oral midazolam at a dose of 0.6 mg/kg prior to dental procedures. Sedative and amnesic effects, patient cooperation, and safety outcomes are assessed and compared to the lower dose group.
  Interventions: Drug: Oral midazolam

INTERVENTIONS:
Drug: Oral midazolam — The intravenous formulation Midazolam Braun 5 mg/ml (B. Braun Melsungen AG, Germany) diluted and mixed with orange juice for oral administration at doses of 0.3 mg/kg , administered approximately 30 minutes before pediatric dental procedures. Sedation and amnesic effects, behavioral cooperation during treatment, sedation onset time, vital signs, recovery duration, safety, and adverse events are systematically monitored and compared between the two dosing groups.
  Arms: Arm 1: Oral Midazolam 0.3 mg/kg
Drug: Oral midazolam — The intravenous formulation Midazolam Braun 5 mg/ml (B. Braun Melsungen AG, Germany) diluted and mixed with orange juice for oral administration at doses of 0.6 mg/kg, administered approximately 30 minutes before pediatric dental procedures. Sedation and amnesic effects, behavioral cooperation during treatment, sedation onset time, vital signs, recovery duration, safety, and adverse events are systematically monitored and compared between the two dosing groups.
  Arms: Arm 2: Oral Midazolam 0.6 mg/kg

SUMMARY:
Dental anxiety frequently impedes effective dental care in pediatric patients. This study aimed to compare the efficacy and safety of two doses (0.3 mg/kg and 0.6 mg/kg) of oral midazolam for sedation and amnesia in preschool children undergoing dental procedures. Methods: This prospective, double-blind, randomized controlled trial included 80 children aged 3-6 years with dental anxiety. Participants were randomly assigned to receive oral midazolam at either 0.3 mg/kg or 0.6 mg/kg. Sedation efficacy, onset time, procedure duration, cooperation level (Houpt Behavior Rating Scale), recovery time, amnesia at 12 hours, 24 hours, and one week, as well as adverse events, were recorded and analyzed

DETAILED DESCRIPTION:
Dental anxiety is common among preschool-aged children, with prevalence rates ranging from 36.5% to 70%. Untreated anxiety often leads to delayed dental care, increased dental caries, and worsened oral health, negatively impacting children and their families. Behavioral management techniques, such as positive reinforcement, are typically employed but may be insufficient for severely anxious patients. Pharmacological sedation, especially with midazolam-a short-acting benzodiazepine-is commonly used to enhance cooperation by providing sedation, anxiety relief, and amnesia. Oral midazolam administration is widely preferred for children due to its non-invasive nature, despite slower onset and variable bioavailability. Current guidelines recommend oral midazolam doses between 0.25 and 1 mg/kg; however, optimal dosing balancing effectiveness and safety remains unclear.

Recognizing this gap, this randomized controlled trial aims to compare two oral midazolam doses (0.3 mg/kg versus 0.6 mg/kg) in preschool children aged 3-6 years who exhibit dental anxiety. Conducted from June to December 2024 at the National Hospital of Odonto-Stomatology in Hanoi, Vietnam, this prospective, double-blind study enrolls 80 pediatric patients who meet strict inclusion and exclusion criteria. Children included have significant dental anxiety, assessed as "negative" or "definitely negative" based on the Frankl Behavior Rating Scale, normal body weight, and an ASA (American Society of Anesthesiologists) physical status of I or II. Patients with systemic diseases, cognitive impairments, severe respiratory conditions, liver or kidney dysfunction, mental disorders (e.g., autism, ADHD), or allergies to sedatives are excluded from participation.

Participants are randomly assigned using block randomization into two groups receiving either 0.3 mg/kg or 0.6 mg/kg oral midazolam. Blinding ensures dentists performing procedures and data collectors remain unaware of dosing specifics to minimize bias. Sedation effectiveness is measured using the Ramsay Sedation Scale (RSS), with successful sedation defined as achieving RSS score 3 ("awake but responds to commands only") within 30 minutes post-administration. Children not reaching this sedation level within the specified timeframe are excluded from further analysis.

Vital signs, including heart rate and oxygen saturation, are closely monitored throughout the procedure. Patient behavior during dental treatment is assessed using the Houpt Behavior Rating Scale, which evaluates sleepiness, movement, and crying. The study also investigates midazolam's amnesic effects through structured memory assessments conducted 12 hours, 24 hours, and one week post-procedure.

Additionally, safety assessments monitor adverse events such as respiratory depression, hypotension, excessive sedation, nausea, and vomiting during sedation and 24 hours afterward. The collected data undergo statistical analysis using SPSS software, employing independent t-tests for continuous variables (e.g., sedation onset time, treatment duration, recovery time) and chi-square or Fisher's exact tests for categorical variables (e.g., sedation success rates, amnesia outcomes). A significance threshold is established at p<0.05.

Through detailed evaluation of sedation efficacy, amnesic effect, patient safety, and procedural cooperation, this research seeks to clarify optimal midazolam dosing strategies, contributing to improved clinical practices, reduced dental anxiety, and better overall pediatric dental experiences.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 3 to 6 years.
* Diagnosed with dental anxiety classified as "definitely negative" or "negative" based on the Frankl Behavior Rating Scale.
* Normal weight range.
* Classified as ASA I or ASA II (American Society of Anesthesiologists Physical Status Classification).

Exclusion Criteria:

* Endocrine disorders, severe respiratory diseases, or heart diseases.
* Mental health conditions such as autism, ADHD, or schizophrenia.
* Abnormal brain development or cognitive impairments.
* Liver or kidney dysfunction.
* Known allergies to benzodiazepines, opiates, etomidate, propofol, ketamine, or other medications used in the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Sedation Effectiveness | Within 30 minutes after oral midazolam administration
  Sedation effectiveness is measured using the Ramsay Sedation Scale (RSS), a standardized 6-point scale evaluating sedation depth. Successful sedation is defined as achieving an RSS score of 3 (awake but responds to commands only) within 30 minutes after administration of oral midazolam. Children not reaching RSS score ≥3 within 30 minutes are classified as having unsuccessful sedation.
Amnesic Effectiveness (Memory Assessment) | 12 hours, 24 hours, and 1 week after the dental procedure
  The ability of pediatric patients to recall details of the dental procedure will be assessed through a structured verbal questionnaire conducted via video call at 12 hours, 24 hours, and one week post-procedure. The assessment aims to determine and compare the amnesic effects between two oral midazolam doses (0.3 mg/kg vs. 0.6 mg/kg)

SECONDARY OUTCOMES:
Sedation Onset Time | Up to 30 minutes after drug administration
  The interval (minutes) from administration of oral midazolam to achieving a sedation score of 3 on the Ramsay Sedation Scale
Patient Behavior During Dental Procedure | During the dental procedure
  Behavior of pediatric patients during the dental procedure will be assessed using the Houpt Behavior Rating Scale, evaluating levels of sleepiness, movement, crying, and overall cooperation. Ratings range from 1 (aborted) to 6 (excellent cooperation).
Recovery Time (PADSS ≥9) | Immediately following procedure until PADSS score ≥9 is achieved
  Recovery time measured from completion of the dental procedure until patients achieve a Post-Anesthetic Discharge Scoring System (PADSS) score of 9 or higher.
Safety and Adverse Events | During the procedure and within 24 hours post-procedure
  Incidence and severity of adverse events, including respiratory depression, hypotension, nausea, vomiting, or excessive sedation occurring during and up to 24 hours post-sedation.
Vital Signs Monitoring | Baseline (T0), immediately after administration (T1), 5 minutes (T2), 10 minutes (T3), 20 minutes (T4), and post-procedure (T5)
  Heart rate and peripheral oxygen saturation (SpO₂) will be monitored and recorded at baseline (pre-sedation, T0), immediately after midazolam administration (T1), and subsequently at intervals of 5 minutes (T2), 10 minutes (T3), 20 minutes (T4), and post-dental procedure (T5), to evaluate safety and physiological response to sedation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical Univeristy, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No